CLINICAL TRIAL: NCT06715917
Title: PROSPECTIVE, MULTICENTRE POST-MARKETING SURVEILLANCE STUDY to ASSESS PERFORMANCE of the GMK UNI ANATOMICAL CEMENTLESS IMPLANT
Brief Title: Multicentre GMK UNI Anatomical Cementless Study - FR
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P02.018.02
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis of the Knee; Avascular Necrosis of the Femoral Condyle; Revision Surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Unicompartmental Knee Arthroplasty (UKA) is the principal surgical alternative to Total Knee Arthroplasty (TKA) in patients with end-stage unicompartmental tibiofemoral osteoarthritis (OA) of the knee. The current post-marketing surveillance study aims to monitor GMK-UNI monocompartmental knee prosthesis performances over a 10-year time period.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with disease that meets the indications for use for Medacta implants included in this study (on-label use);
* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to the patient's surgery;
* Patient's age between 18 and 75 years old;
* Patients must be willing to comply with the pre and postoperative evaluation schedule.

Exclusion Criteria:

* Patients with one or more medical conditions identified as a contraindication defined by the labelling on any Medacta implants used in this study;
* Any patient who cannot or will not provide informed consent for participation in the study;
* Patients who need a revision surgery
* Patients unable to understand and take action;
* Any case not described in the inclusion criteria;
* Patients aged under 18 years;
* Patients aged over 75 years;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion/exclusion criteria to take part to the current clinical study will be invited to participate before the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2032-03-06 (Estimated); Study Completion 2032-03-06 (Estimated)

PRIMARY OUTCOMES:
New Knee Society Score (KSS) | Preoperative, 3 months, 1, 2, 3, 5, 7 and 10 years
  The new Knee Society Knee Scoring System is both physician and patient derived. It includes versions to be administered preoperatively and postoperatively. It has an initial assessment of demographic details, including an expanded Charnley functional classification. The objective knee score, completed by the surgeon, includes a VAS score of pain walking on level ground and on stairs or inclines, as well as an assessment of alignment, ligament stability, and ROM, along with deductions for flexion contracture or extensor lag. Patients then record their satisfaction, functional activities, and expectations. Given the diverse activity profiles of many contemporary patients, the functional component of the score was improved to include a patient-specific survey, which evaluates features such as standard activities of daily living, patient-specific sports and recreational activities, patient satisfaction, and patient expectations

SECONDARY OUTCOMES:
Kujala Score | 3 months, 1, 2, 3, 5, 7 and 10 years
  The "Kujala Score" is the eponymous name for the Anterior Knee Pain Scale (AKPS). It is a patient-reported outcome survey and diagnostic tool that aims to assess the severity of symptoms and physical limitations in patients with patellofemoral pain syndrome (PFPS). The Kujala Score is a self-administered questionnaire for PFPS patients consisting of 13 questions that relate to specified activities, pain severity, and clinical symptoms. It is scored out of 100 points, which represents the summation of the scores for each individual question
Survival of the implant | 3 months, 1, 2, 3, 5, 7 and 10 years
  Survival rate assessed with Kaplan Meier analysis
Safety of the implant | Intraoperative, 3 months, 1, 2, 3, 5, 7 and 10 years
  Recording of any adverse event and complication (including but not limited to: infection, loosening, deep venous thrombosis (DVT), fracture, reflex sympathetic dystrophy syndrome (RSD).)

CONTACTS AND LOCATIONS:
Locations (5):
- France (4):
  - Clinique Saint Vincent de Paul, Bourgoin
  - Polyclinique du Parc, Caen
  - Clinique du Mail, La Rochelle
  - Centre Orthéo, Saint-Etienne
- Bürgerspital Solothurn, Solothurn, Switzerland